CLINICAL TRIAL: NCT03534934
Title: CT-Based Modeling of Bone Micro-Architecture and Fracture-Risk in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Punam K Saha (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Punam K Saha, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 201802724; R01HL142042 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-05-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Osteoporosis
Keywords: COPD; Osteoporosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Osteoporosis | interventions — Vital Signs; Surveys and Questionnaires; Hematologic Tests; Absorptiometry, Photon; Multidetector Computed Tomography; Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: All subjects will participate in both baseline and three year follow-up visits and undergo identical interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Baseline (Experimental): Smokers, defined has having at least a 10 pack-year lifetime history, with and without COPD will participate in the following interventions:
  Vital Signs Urine Pregnancy Test on woman of child bearing potential Pre- and Post-Bronchodilator Spirometry Questionnaires Blood Test for Vitamin D level, Hemoglobin A1c, and creatinine level Duel-energy X-ray absorptiometry scan (DXA) of the whole body, spine, and hip Duel-energy X-ray absorptiometry scan (DXA) for vertebral fracture assessment Multi-detector computed tomography (MDCT) of the hip and ankle
  Interventions: Diagnostic Test: Vital signs; Diagnostic Test: Urine Pregnancy Test; Other: Questionnaires; Diagnostic Test: Blood Test; Diagnostic Test: Duel-energy X-ray absorptiometry scan; Diagnostic Test: Multi-detector computed tomography; Diagnostic Test: Dual-energy X-ray absorptiometry scan
- 3 year follow-up (Experimental): All subjects who completed a baseline visit will return for a follow-up visit and participate in the following interventions:
  Vital Signs Urine Pregnancy Test on woman of child bearing potential Pre- and Post-Bronchodilator Spirometry Questionnaires Blood Test for Vitamin D level, Hemoglobin A1c, and creatinine level Duel-energy X-ray absorptiometry scan (DXA) of the whole body, spine, and hip Duel-energy X-ray absorptiometry scan (DXA) for vertebral fracture assessment Multi-detector computed tomography (MDCT) of the hip and ankle
  Interventions: Diagnostic Test: Vital signs; Diagnostic Test: Urine Pregnancy Test; Other: Questionnaires; Diagnostic Test: Blood Test; Diagnostic Test: Duel-energy X-ray absorptiometry scan; Diagnostic Test: Multi-detector computed tomography; Diagnostic Test: Dual-energy X-ray absorptiometry scan

INTERVENTIONS:
Diagnostic Test: Vital signs — Heart rate, respirations, blood pressure, temperature, oxygen saturation
  arterial oxygen saturation (SaO2), height and weight
Diagnostic Test: Urine Pregnancy Test — Urine pregnancy test done on woman of childbearing potential.
Other: Questionnaires — Subject Questionnaire Calcium Intake Questionnaire Home and Work Activities Survey
Diagnostic Test: Blood Test — Blood test for vitamin D level, Hemoglobin A1c, and creatinine level
Diagnostic Test: Duel-energy X-ray absorptiometry scan — Bone density measurement
  Other Names: DXA scan
Diagnostic Test: Multi-detector computed tomography — Hip and ankle CT scan
  Other Names: MDCT, CT scan
Diagnostic Test: Dual-energy X-ray absorptiometry scan — Vertebral fracture assessment
  Other Names: DXA scan

SUMMARY:
The goal of this translational study is to establish a newly emerging CT-based tool for the characterization of changes in bone micro-architecture and assessment of their implications for fracture-risk in a population of COPD patients at risk for osteoporosis. The tool will be suitable and generalizable across emerging CT scanners from different vendors, and it will provide a more structurally-based assessment of osteoporosis and bone loss than is provided by simple bone density measures. The study will characterize the impact of different COPD-related factors on bone structure, and their implications for fracture-risk, leading to the development of a COPD-specific model for assessment of fracture-risk that will utilize patient-specific demographic, clinical and radiographic data, and CT BMD at the spine, as well as bone structural measures at the hip and/or ankle.

DETAILED DESCRIPTION:
This translational study seeks to establish a Chronic Obstructive Pulmonary Disease (COPD)-specific fracture prediction model using the investigators unique computed tomography (CT)-based assessment of peripheral bone micro-architecture. Osteoporosis, a common comorbidity among patients with COPD, accelerates morbidity and mortality. The basis for this comorbidity is poorly understood, thus the need for characterizing the link between COPD-related factors and bone micro-architecture and their association to fracture-risk. Multiple COPD-related factors are associated with osteoporosis. Different COPD-related causes of bone loss may non-uniformly impact cortical and trabecular bone structures with varying mechanical consequences, reflective of divergent COPD-associated fracture-risk in individuals with similar bone mineral density (BMD). Little is known about this linkage, and the study goal is to fill this knowledge gap using a clinically suitable emerging CT-based tool for characterization of bone micro-architecture at peripheral sites. Specifically, this study will-(1) establish the generalizability of the investigators bone micro-architecture assessment applied to emerging low dose / high resolution CT scanners from different vendors; (2) assess its potential as compared to dual energy x-ray absorptiometry (DXA) to explain prevalent fractures and predict incident fractures among patients with COPD; (3) quantify the impact of different COPD-related factors on bone structures and their implications for fracture-risk; (4) identify COPD subtypes with rapid bone structural degeneration; and (5) develop a COPD-specific model for assessment of fracture-risk using patient-specific data.

The study will take advantage of-(1) existing COPD patient cohorts with lung characterization at the University of Iowa (UI) and Columbia University (CU) representing a wide demographic range; (2) access to emerging CT scanners at both sites; and (3) unique image processing methodologies for quantifying three-dimensional bone structural metrics. The study will recruit 550 smokers with and without COPD from the UI and CU cohorts of the COPDGene and SPIROMICS studies. Smokers without COPD will comprise the control group for the study. At baseline and 3-year follow-up visits, the study team will collect-(1) data related to risk factors; (2) a lateral spine CT scout scan to assess vertebral fractures; (3) high resolution CT scans of the hip and ankle for computation of bone structural metrics; (4) whole-body, spine and hip DXA scans for evaluation of bone mineral density and body composition; and (5) DXA vertebral fracture assessment.

This study will establish an emerging CT-based scanner-independent generalizable tool to assess bone response to different therapeutic interventions aimed at slowing or reversing bone loss, and possibly restoring bone structure, potentially leading to more patient-specific interventions. Also, this study seeks to explain the relationships among various COPD-related factors, bone structural changes and their implications for fracture-risk.

Finally, a COPD-specific model for assessment of fracture-risk will be developed that will utilize patient-specific demographic, clinical and radiographic data, and CT BMD at the spine, as well as bone structural measures at the hip and/or ankle.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smoker, defined as having at least 10-pack year lifetime history
* Age: 45-90

Subjects will be stratified into groups based on COPD disease status: smokers with COPD and smokers without COPD.

Smokers with COPD will be further stratified into three groups: low emphysema (< 3%), moderate emphysema (between 3 and 10%), and severe emphysema (> 10%).

Exclusion Criteria:

* Pregnant or breast-feeding
* Metastatic Malignancy
* Currently receiving dialysis
* Any lower extremity fracture within the last year
* Any lower extremity fracture with hardware implant(s)
* History of bilateral tibia fractures

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Prevalent vertebral fractures at baseline | Baseline Visit
  Method: Prevalent fracture cases at the baseline visit will be determined using expert visual reading of the baseline lateral spine CT scout scan.
CT-based fracture-risk | Baseline Visit
  Method: Fragility fracture-risk will be computed using a CT-based model comprising of patient-specific demographic, clinical and radiographic data, CT bone mineral density at the spine, and CT bone micro-structural measures at the ankle.
DXA-based fracture risk | Baseline Visit
  Method: Fragility fracture-risk will be computed using a DXA-based model comprising of patient-specific demographic, clinical and radiographic data, and whole-body, spine, and hip DXA bone mineral density.

SECONDARY OUTCOMES:
CT bone mineral density at the spine | Change from baseline and three year follow up visit
  Method: CT measures of thoracic spine bone mineral density will be computed using a chest CT scan and computerized algorithms.
DXA Bone Mineral Density | Change from baseline and three year follow up visit.
  DXA Bone Mineral Density score will be obtained using standard DXA scans.

CONTACTS AND LOCATIONS:
Overall Officials: Punam Saha, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Clinical exam, questionnaire, and image-derived data will be made available to other researchers who request it formally. The data will be de-identified and linked only by code numbers. To further minimize the risk of breaches of confidentiality, we will establish data-use sharing agreements, and consider employment of electronic firewalls, locked storage facilities, password authentication of users, audit trails, and disaster prevention/recovery plans. We will stipulate that data are used only for research purposes, that proposed research using the data will be reviewed by an Institutional Review Board, and data will not be transferred to other users. The data would be available upon completion of necessary data management and statistical analyses. At that time, data could be provided on appropriate storage media via mail. Data files would be provided in SAS format, with PDF documentation files. We also will provide copies of questionnaires and images from which our data are derived.
Time Frame: The data would be available about 12 months after completion of the grant, with necessary data management and statistical analyses done by then. At that time, data could be provided on the appropriate storage media through the mail, with appropriate variable labels and other necessary documentation.
Access Criteria: Data will only be available to researchers who formally request it and who have entered into a data-use agreement with the principal investigators.